CLINICAL TRIAL: NCT02149316
Title: Cardioprotective Effects of Remote Ischemic Preconditioning With Postconditioning of the Recipient on Donor Heart in Heart Transplantation Surgery
Brief Title: Remote Ischemic Preconditioning With Postconditioning in Heart Transplantation Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Guyan Wang, The Chief of Infection-Control Department, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FW2012-863B-C
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Myocardial Ischemic Reperfusion Injury; End Stage Heart Disease; Heart Failure; Cardiomyopathy
MeSH Terms: conditions — Myocardial Reperfusion Injury; Heart Failure; Cardiomyopathies

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RIPC+RIPostC (Experimental)
  Interventions: Procedure: RIPC+RIPostC
- control (Sham Comparator)
  Interventions: Procedure: control

INTERVENTIONS:
Procedure: RIPC+RIPostC — Four 5 min cycles of upper limb ischemia and reperfusion by a cuff inflated to 200 mmHg, twice (after anesthesia induction and before surgery started, at 20min after aortic declamping)
  Arms: RIPC+RIPostC
Procedure: control — a deflated cuff placed on the right upper arm
  Arms: control

SUMMARY:
The purpose of this study is to determine whether remote ischemic preconditioning with postconditioning (RIPC+RIPostC) reduces myocardial injury and improves clinical outcomes in heart transplantation surgery.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective orthotopic heart transplantation surgery

Exclusion Criteria:

* peripheral vascular disease affecting the upper arms
* mechanical circulatory support before surgery
* taking the antidiabetic sulphonylurea, glibenclamide
* cold ischemic time of donor heart > 12 hours
* repeated heart surgery

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
serum cardiac troponin I (cTnI) | within 72 hours after aortic declamping

SECONDARY OUTCOMES:
plasma microRNA-133b (miR-133b) | within 72 hours after aortic declamping
plasma microRNA-208a (miR-208a) | within 72 hours after aortic declamping

CONTACTS AND LOCATIONS:
Overall Officials: Guyan Wang, PhD, Principal Investigator — State Key Laboratory of Cardiovascular Disease, Fuwai Hospital, National Center for Cardiovascular Diseases, CAMS and PUMC, Beijing, China
Locations (1):
- State Key Laboratory of Cardiovascular Disease, Fuwai Hospital, National Center for Cardiovascular Diseases, CAMS and PUMC, Beijing, China